CLINICAL TRIAL: NCT05527795
Title: Predictive Clinical Features for Response to Adjuvant Immunotherapy in Stage II,III and IV Resected Melanoma
Acronym: Mel-ImmAdj
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 616
Record Dates: First submitted 2022-05-17; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: Melanoma; adjuvant immunotherapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-mutated: Non mutated (BRAF or NRAS) stage II, III or IV (resected) melanoma patients treated with first line adjuvant immunotherapy (anti-PD-1 with either pembrolizumab or nivolumab)
  Interventions: Other: Frequency and duration of response to adjuvant immunotherapy according to clinical features; Other: Frequency of each type of relapse (i. e. local, distant, unique or multiple) to adjuvant therapy according to clinical features; Other: Duration of relapse-free survival according to clinical features; Other: Duration of overall survival according to clinical features; Other: Overall response rate; Other: Frequency of adverse events according to clinical features
- BRAF-mutated: BRAF-mutated stage II, III or IV (resected) melanoma patients treated with first line adjuvant immunotherapy (anti-PD-1 with either pembrolizumab or nivolumab)
  Interventions: Other: Frequency and duration of response to adjuvant immunotherapy according to clinical features; Other: Frequency of each type of relapse (i. e. local, distant, unique or multiple) to adjuvant therapy according to clinical features; Other: Duration of relapse-free survival according to clinical features; Other: Duration of overall survival according to clinical features; Other: Overall response rate; Other: Frequency of adverse events according to clinical features
- NRAS-mutated: NRAS-mutated (BRAF or NRAS) stage II, III or IV (resected) melanoma patients treated with first line adjuvant immunotherapy (anti-PD-1 with either pembrolizumab or nivolumab)
  Interventions: Other: Frequency and duration of response to adjuvant immunotherapy according to clinical features; Other: Frequency of each type of relapse (i. e. local, distant, unique or multiple) to adjuvant therapy according to clinical features; Other: Duration of relapse-free survival according to clinical features; Other: Duration of overall survival according to clinical features; Other: Overall response rate; Other: Frequency of adverse events according to clinical features

INTERVENTIONS:
Other: Frequency and duration of response to adjuvant immunotherapy according to clinical features — * Frequency of relapse to adjuvant immunotherapy according to clinical features
  * Duration of relapse as defined by the time (days) between adjuvant immunotherapy onset and relapse date according to clinical features
Other: Frequency of each type of relapse (i. e. local, distant, unique or multiple) to adjuvant therapy according to clinical features — Percentages of each type of relapse (i. e. local, distant, unique or multiple) according to clinical features
Other: Duration of relapse-free survival according to clinical features — Duration of relapse-free survival as defined by the time (days) between adjuvant immunotherapy onset and relapse date.
Other: Duration of overall survival according to clinical features — Duration of relapse-free survival as defined by the time (days) between adjuvant immunotherapy onset and the date of death (irrespectively of the cause) 10 years after inclusion in the study. Alive or lost to follow-up patients will be censored at the date of the last follow-up visit.
Other: Overall response rate — Response rate to adjuvant immunotherapy and to treatment lines subsequent to relapse. Response rate to adjuvant immunotherapy is defined by the absence of relapse as assessed by the physician following the first year of adjuvant therapy. Response to treatment after relapse is defined as partial or complete response as assessed by the physician following the first year of adjuvant therapy.
Other: Frequency of adverse events according to clinical features — Rate of adverse events according to their nature and grade (as defined by CTCAE V 5.0) and according to clinical features

SUMMARY:
Surgical excision is the treatment of choice for stage II, III and resectable stage IV melanoma and is curative in most cases. Given the recent success of immunotherapy for the treatment of patients with advanced metastatic melanoma, the use of immunotherapy has been evaluated in the adjuvant setting for patients at high risk of recurrence. In this context, Nivolumab prolonged Recurrence-Free Survival (RFS) while reducing toxicity compared with Ipilimumab in a phase III clinical trial, and was subsequently FDA-approved in December 2017 for adjuvant treatment of locally advanced melanoma with metastatic lymph node involvement after resection of cutaneous lesions. While a fraction of patients benefit from adjuvant PD-1 immunotherapy, approximately 40% of patients are still relapsing despite this adjuvant treatment, without being able to identify them early and with poor understanding of resistance mechanisms. Additionally, about 15% of the patients will develop serious adverse effects driven by immunotherapy and often discontinuing or even contraindicating the onset of subsequent treatments, hence affecting global patients care. It is therefore of prime importance to identify clinical features able to predict response and toxicities to adjuvant immunotherapy in melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage II, III or IV (resected) melanoma
* Treated by surgery and adjuvant immunotherapy between January 1st of 2019 and January 1st of 2029
* Gave informed consent to allow the use of biological samples for research purpose
* Has read the information sheet regarding this study
* With tumor samples available at the biobank center

Exclusion Criteria:

* Patients under 18 years old
* Patients placed under the judicial protection
* Opposed to this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stage II, III and IV (resected) melanoma patients treated with surgery and adjuvant immunotherapy in the dermatology unit of Lyon-Sud hospital between January 1st of 2019 and January 1st of 2029, with no residual disease prior to immunotherapy onset.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2039-01-01 (Estimated)

PRIMARY OUTCOMES:
Duration of response to adjuvant immunotherapy according to clinical features. | 1 year
  • Duration of response as defined by the time (days) between adjuvant immunotherapy onset and relapse date according to clinical features.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No